CLINICAL TRIAL: NCT02392078
Title: Laser Ablation of Abnormal Neurological Tissue Using Robotic NeuroBlate System (LAANTERN) Prospective Registry
Brief Title: Laser Ablation of Abnormal Neurological Tissue Using Robotic NeuroBlate System
Acronym: LAANTERN
Status: Completed | Type: Observational
Sponsor: Monteris Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: LAANTERN
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Brain Tumor; Primary Brain Tumor; Epileptic/Seizure Foci; Movement Disorders
Keywords: Procedural Success; Progression; Quality of Life; Seizure Freedom; Progression Free Survival; Overall Survival
MeSH Terms: conditions — Brain Neoplasms; Epilepsy; Movement Disorders; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: NeuroBlate System

SUMMARY:
The NeuroBlate® System (NBS) is a minimally invasive robotic laser thermotherapy tool that is being manufactured by Monteris Medical. Since it received FDA clearance in May 2009, the NBS has been used in over 2600 procedures conducted at over 70 leading institutions across United States. This is a prospective, multi-center registry that will include data collection up to 5 years to evaluate safety, QoL, and procedural outcomes including local control failure rate, progression free survival, overall survival, and seizure freedom in up to 3,000 patients and up to 50 sites.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or legally authorized representative provides written authorization and/or consent
2. Subject who is to undergo thermal therapy by the NeuroBlate® System for treatment of their neurological disorder

Exclusion Criteria:

1. Subject who is, or is expected to be inaccessible for follow-up
2. Other concurrent medical or other condition (chronic or acute in nature) that in the opinion of the investigator, may prevent participation or otherwise render subject ineligibility for the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who present with a brain lesion, epileptic/seizure foci, or movement disorder who have been deemed appropriate candidates, in the opinion of the treating physician, for laser ablation using the NeuroBlate® System.
Sampling Method: Non-Probability Sample
Enrollment: 1153 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Leuthardt, MD, Principal Investigator — Washington University School of Medicine
Locations (26):
- United States (26):
  - Barrow Neurological Institute at Dignity Health St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California, San Diego, La Jolla, California
  - Children's Hospital of Orange County, Orange, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Advent Health Orlando, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - The Cleveland Clinic Florida, Weston, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - University of Minnesota, Minneapolis, Minnesota
  - United Children's Hospital St. Paul, Saint Paul, Minnesota
  - Washington University, St Louis, Missouri
  - New York University Langone Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Saint Thomas West Hospital and Research Institute, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson, Houston, Texas

REFERENCES:
- [Derived] Landazuri P, Shih J, Leuthardt E, Ben-Haim S, Neimat J, Tovar-Spinoza Z, Chiang V, Spencer D, Sun D, Fecci P, Baumgartner J. A prospective multicenter study of laser ablation for drug resistant epilepsy - One year outcomes. Epilepsy Res. 2020 Nov;167:106473. doi: 10.1016/j.eplepsyres.2020.106473. Epub 2020 Sep 22. PMID 33045664
- [Derived] Kim AH, Tatter S, Rao G, Prabhu S, Chen C, Fecci P, Chiang V, Smith K, Williams BJ, Mohammadi AM, Judy K, Sloan A, Tovar-Spinoza Z, Baumgartner J, Hadjipanayis C, Leuthardt EC. Laser Ablation of Abnormal Neurological Tissue Using Robotic NeuroBlate System (LAANTERN): 12-Month Outcomes and Quality of Life After Brain Tumor Ablation. Neurosurgery. 2020 Sep 1;87(3):E338-E346. doi: 10.1093/neuros/nyaa071. PMID 32315434
- [Derived] Rennert RC, Khan U, Bartek J, Tatter SB, Field M, Toyota B, Fecci PE, Judy K, Mohammadi AM, Landazuri P, Sloan AE, Kim AH, Leuthardt EC, Chen CC. Laser Ablation of Abnormal Neurological Tissue Using Robotic Neuroblate System (LAANTERN): Procedural Safety and Hospitalization. Neurosurgery. 2020 Apr 1;86(4):538-547. doi: 10.1093/neuros/nyz141. PMID 31076762

RESULTS

PARTICIPANT FLOW:
Groups:
- Metastatic Brain Tumor: All eligible study subjects who presented with a metastatic brain tumor.
- Primary Brain Tumor: All eligible study subjects who presented with a primary brain tumor.
- Epileptic/Seizure Foci: All eligible study subjects who presented with epilepsy or seizure foci.
- Movement Disorders: All eligible study subjects who presented with a movement disorder.
Period: Overall Study
Arm/Group | Metastatic Brain Tumor | Primary Brain Tumor | Epileptic/Seizure Foci | Movement Disorders
Started | 374 | 488 | 288 | 3
Completed | 342 | 445 | 268 | 2
Not Completed | 32 | 43 | 20 | 1
Not completed — Did not have procedure | 32 | 43 | 20 | 1

BASELINE CHARACTERISTICS:
Population: 1057 subjects total across 4 cohorts- 268 Epilepsy, 2 Movement disorders, 445 Primary brain tumors and 342 Metastatic brain tumors for a total of 1057.
Groups:
- Metastatic Tumor: All eligible study subjects who presented with a metastatic brain tumor.
- Primary Tumor: All eligible study subjects who presented with a primary brain tumor.
- Epilepsy: All eligible study subjects who presented with epilepsy or seizure foci.
- Movement Disorder: All eligible study subjects who presented with a movement disorder.
- Total: Total of all reporting groups
Arm/Group | Metastatic Tumor | Primary Tumor | Epilepsy | Movement Disorder | Total
Number analyzed (Participants) | 342 | 445 | 268 | 2 | 1057
Age, Customized [Median (Full Range); unit: years] | 61.9 [21.6 to 95.8] | 53.7 [6.6 to 87] | 33.9 [2.5 to 72.3] | 66.9 [57.4 to 75.6] | 54.7 [2.5 to 95.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 205 | 191 | 139 | 1 | 536
  Male | 137 | 254 | 129 | 1 | 521
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 23 | 37 | 0 | 74
  Not Hispanic or Latino | 325 | 416 | 225 | 2 | 968
  Unknown or Not Reported | 3 | 6 | 6 | 0 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 2
  Asian | 4 | 9 | 5 | 0 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 39 | 19 | 21 | 0 | 79
  White | 288 | 406 | 222 | 2 | 918
  More than one race | 2 | 1 | 5 | 0 | 8
  Unknown or Not Reported | 8 | 9 | 15 | 0 | 32
Region of Enrollment [Number; unit: participants]
  United States | 342 | 445 | 268 | 2 | 1057

OUTCOME MEASURES:

1. Primary Outcome: Safety (Reportable Adverse Events)
Description: Safety profile described by the NBS and surgical-related AEs
Time Frame: up to 5 years or last follow up
Measure: Count of Participants; unit: Participants
Groups:
- Number of Participants: All eligible study subjects who underwent LITT with the NeuroBlate System.
Arm/Group | Number of Participants
Number analyzed (Participants) | 1057
Participants
  Anxiety | 1
  Aphasia | 7
  Ataxia or loss of body coordination | 2
  Bleeding or increased risk of bleeding into or around the brain | 30
  Blurry vision/visual disturbance/Permanent neuro deficit | 3
  Cerebral edema/Edema | 21
  Cerebral infarction | 1
  Complete or incomplete hemiparesis | 2
  Deep venous thrombsois | 2
  Difficulty speaking | 5
  Difficulty walking | 3
  Headache | 3
  Infection or increased risk of infection, local or generalized | 6
  Injury to brain tissue | 2
  Muscle weakness | 15
  Nausea/vomiting | 1
  Nerve Paralysis/Paralysis | 3
  Personality or cognitive changes (e.g. mood, memory, attention and thinking ability) | 3
  Pneumonia | 3
  Pulmonary or other air embolism | 7
  Seizure/Increased seizures frequency, duration or severity | 19
  Status epilepticus | 1
  Stroke or transient ischemic attack (TIA) | 2
  Tingling or numb sensations in the body | 1
  Wound dehiscence | 2
  Other | 23
  Hypertension | 1
  None | 888

2. Primary Outcome: Reason for NeuroBlate
Description: To identify the primary reason the NeuroBlate system was chosen for subject
Time Frame: Index procedure
Measure: Number; unit: participants
Groups:
- Subjects Treated With NeuroBlate LITT: All eligible study subjects who underwent LITT with the NeuroBlate System.
Arm/Group | Subjects Treated With NeuroBlate LITT
Number analyzed (Participants) | 1057
participants
  Minimally Invasive Preferred | 702
  Non-Resectable | 186
  Subject exceeded max dose or could not tolerate radiation | 24
  Subject not a candidate for craniotomy | 31
  Palliative | 7
  Other | 139
  Unknown | 37

3. Primary Outcome: Number of Patients Demonstrating Seizure Freedom (ENGEL and ILAE Classifications)
Description: Collected for all subjects by disease etiology.
  Seizure freedom assessed for all subjects with epilepsy at time of last follow-up. The ENGEL surgical outcome scale is composed of four classes of epilepsy (Class I (best), Class II, Class III, Class IV (worst)) categorized by severity. The ILAE outcome scale contains six classes (Class 1 (best), 2, 3, 4, 5, 6 (worst)) categorized by severity.
Time Frame: up to 5 years or last follow up
Population: Data not collected for various cohorts because they were not applicable to the end points associated with those cohorts disease state.
Measure: Count of Participants; unit: Participants
Arm/Group | Metastatic Brain Tumor | Primary Brain Tumor | Epileptic/Seizure Foci | Movement Disorders
Number analyzed (Participants) | 342 | 445 | 268 | 2
Participants
  ENGEL I: number analyzed (Participants) | 0 | 0 | 268 | 0
  ENGEL I |  |  | 88 |
  ENGEL II: number analyzed (Participants) | 0 | 0 | 268 | 0
  ENGEL II |  |  | 34 |
  ENGEL III: number analyzed (Participants) | 0 | 0 | 268 | 0
  ENGEL III |  |  | 29 |
  ENGEL IV: number analyzed (Participants) | 0 | 0 | 268 | 0
  ENGEL IV |  |  | 21 |
  ENGEL Not Provided: number analyzed (Participants) | 0 | 0 | 268 | 0
  ENGEL Not Provided |  |  | 96 |
  ILAE 1: number analyzed (Participants) | 0 | 0 | 268 | 0
  ILAE 1 |  |  | 58 |
  ILAE 2: number analyzed (Participants) | 0 | 0 | 268 | 0
  ILAE 2 |  |  | 25 |
  ILAE 3: number analyzed (Participants) | 0 | 0 | 268 | 0
  ILAE 3 |  |  | 31 |
  ILAE 4: number analyzed (Participants) | 0 | 0 | 268 | 0
  ILAE 4 |  |  | 36 |
  ILAE 5: number analyzed (Participants) | 0 | 0 | 268 | 0
  ILAE 5 |  |  | 16 |
  ILAE 6: number analyzed (Participants) | 0 | 0 | 268 | 0
  ILAE 6 |  |  | 4 |
  ILAE Not Provided: number analyzed (Participants) | 0 | 0 | 268 | 0
  ILAE Not Provided |  |  | 98 |

4. Primary Outcome: Change in Quality of Life
Description: Assessed with following questionnaires:
  1. KPS (malignancy subjects only) Scale range 0-100 measuring the ability of patients with cancer to perform ordinary daily activities. Score 0 is dead, 100 is no disease symptoms
  2. FACT-Br (malignancy subjects only) Measure general quality of life across 5 scales- physical well-being, social/family well-being, emotional well-being, functional well-being & other. Higher score, better quality of life. Range 0-200
  3. EQ-5D (tumor/epilepsy subjects only) Measure of health consisting of the descriptive system & the visual analogue scale (VAS). The system assesses subject mobility, self-care, usual activities, pain/discomfort & anxiety/depression. Higher score, better quality of life. Range 0-100
  4. QOLIE-31 (epilepsy subjects only) 7 scales assessing emotional well-being, social functioning, energy/fatigue, cognitive functioning, seizure worry, medication effects, & overall quality of life. Higher score, better quality of life. Range 0-100
Time Frame: up to 5 years or last follow-up
Population: The questionnaires are only applicable to certain cohorts in the study population and were not collected or analyzed for subjects who were not in that cohort.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Metastatic Brain Tumor | Primary Brain Tumor | Epileptic/Seizure Foci | Movement Disorders
Number analyzed (Participants) | 342 | 445 | 268 | 2
score on a scale
  KPS: number analyzed (Participants) | 342 | 445 | 0 | 0
  KPS | 90 [0 to 100] | 80 [10 to 100] |  |
  FACT Br: number analyzed (Participants) | 342 | 445 | 0 | 0
  FACT Br | 149 [49 to 200] | 149 [49 to 200] |  |
  EQ-5D: number analyzed (Participants) | 342 | 445 | 268 | 0
  EQ-5D | 80 [5 to 100] | 80 [5 to 100] | 80 [1 to 100] |
  QOLIE-31: number analyzed (Participants) | 0 | 0 | 268 | 0
  QOLIE-31 |  |  | 65.3 [7 to 96] |

5. Primary Outcome: Number of Patients Demonstrating Local Control and Overall Survival
Description: Collected for all subjects by disease etiology.
  Local control as measured by time to local tumor recurrence.
  Overall survival assessed by Kaplan-Meier method.
Time Frame: up to 5 years or last follow up
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Median (in years)
Arm/Group | Metastatic Brain Tumor | Primary Brain Tumor | Epileptic/Seizure Foci | Movement Disorders
Number analyzed (Participants) | 342 | 445 | 268 | 2
Median (in years)
  Local Control: Median time from procedure to tumor progression (years): number analyzed (Participants) | 342 | 445 | 0 | 0
  Local Control: Median time from procedure to tumor progression (years) | 3.44 [1.7 to NA] — Upper limit is NA due to over half of the subjects still being alive at time of study exit | 3.26 [2.02 to NA] — Upper limit is NA due to over half of the subjects still being alive at time of study exit |  |
  Overall Survival: Median time from diagnosis to death (years): number analyzed (Participants) | 342 | 445 | 0 | 0
  Overall Survival: Median time from diagnosis to death (years) | 4.69 [3.38 to 5.73] | 4.27 [3.68 to 7.34] |  |

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of patient consent (prior to the surgical procedure) to study withdraw/completion which varied for each subject, but up to 5 years. From time of consent to withdraw varied based on death or study withdraw. Adverse events were monitored throughout the subjects study participation.
Groups:
- Number of Participants With Adverse Events: All eligible study subjects who underwent LITT with the NeuroBlate System.
Arm/Group | Number of Participants With Adverse Events
All-Cause Mortality (participants affected / at risk) | 367/1057
Serious Adverse Events (participants affected / at risk) | 31/1057
Other Adverse Events (participants affected / at risk) | 169/1057
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Number of Participants With Adverse Events (N=1057)
Aphasia (Nervous system disorders) | 1 (1)
Bleeding or increased bleeding around the brain (Nervous system disorders) | 7 (7)
Cerebral edema (Nervous system disorders) | 2 (2)
Edema (Blood and lymphatic system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Infection or increased risk of infection (Infections and infestations) | 2 (2)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Nerve paralysis (Nervous system disorders) | 1 (1)
Pulmonary or other air embolism (Cardiac disorders) | 3 (3)
Seizures (Nervous system disorders) | 4 (4)
Status epilepticus (Nervous system disorders) | 1 (1)
Stroke or transient ischemic attack (Cardiac disorders) | 2 (2)
Other (General disorders) | 10 (10)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Number of Participants With Adverse Events (N=1057)
Anxiety (Psychiatric disorders) | 1 (1)
Aphasia (Nervous system disorders) | 7 (7)
Ataxia or loss of body coordination (Nervous system disorders) | 2 (2)
Bleeding or increased risk of bleeding around the brain (Nervous system disorders) | 30 (30)
Blurry vision/visual disturbance (Nervous system disorders) | 3 (3)
Cerebral edema/Edema (Blood and lymphatic system disorders) | 21 (21)
Cerebral infarction (Nervous system disorders) | 1 (1)
Complete or incomplete hemiparesis (Nervous system disorders) | 2 (2)
Deep venous thrombosis (Cardiac disorders) | 2 (2)
Difficulty speaking (Nervous system disorders) | 5 (5)
Difficulty walking (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (3)
Infection or increased risk of infection (Infections and infestations) | 6 (6)
Injury to brain tissue (Nervous system disorders) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 15 (16)
Nausea/vomiting (Gastrointestinal disorders) | 1 (1)
Nerve paralysis/paralysis (Nervous system disorders) | 3 (3)
Personality or cognitive changes (Psychiatric disorders) | 3 (3)
Pneumonia (Infections and infestations) | 3 (3)
Pulmonary or air embolism (Cardiac disorders) | 7 (7)
Seizure/increased seizures frequency, duration, or severity (Nervous system disorders) | 19 (22)
Status epilepticus (Nervous system disorders) | 1 (1)
Stroke or transient ischemic attack (Cardiac disorders) | 2 (2)
Tingling or numb sensations in the body (Nervous system disorders) | 1 (1)
Wound dehiscence (Skin and subcutaneous tissue disorders) | 2 (2)
Other (General disorders) | 23 (25)
Hypertension (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/78/NCT02392078/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT02392078/SAP_001.pdf